CLINICAL TRIAL: NCT00469547
Title: Safety & Acceptance of 62% & 15% Ethanol in Emollient Gel as Topical Male Microbicides
Brief Title: 62% & 15% Ethanol in Emollient Gel as Topical Male Microbicides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: King Holmes, MD, PhD, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 30225-D; KEMRI HSD #SCC931; 06-0040
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Sexually Transmitted Infections
Keywords: ethanol, microbicide, sexually transmitted, Kenya, males; HIV Seronegativity
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 62% ethanol in emollient gel
  Interventions: Other: 62% ethanol in emollient gel
- 2 (Placebo Comparator): 15% ethanol in emollient gel
  Interventions: Drug: Placebo; Other: 15% ethanol in emollient gel

INTERVENTIONS:
Other: 62% ethanol in emollient gel — 62% ethanol in emollient gel used as a topical male microbicide
  Other Names: Topical male microbicide
  Arms: 1
Drug: Placebo — 15% ethanol in emollient gel used as a topical male microbicide
  Other Names: Topical male microbicide
  Arms: 2
Other: 15% ethanol in emollient gel — 15% ethanol in emollient gel used as a topical male microbicide
  Other Names: Topical male microbicide
  Arms: 2

SUMMARY:
The purpose of this study is to look at the safety and acceptance of using a microbicide (product that kills germs) gel to clean the genital area. Microbicide gel is used by hospital workers to clean their hands to kill germs. Researchers hope to use information from this study to conduct a larger study to determine if the microbicidal gel protects men against sexually transmitted infections, including HIV. Thirty healthy uncircumcised Kenyan men, 18 years and older, working in the fishing industry in Kisumu will be recruited. Participants will complete a questionnaire about their background and sexual practices. A researcher will conduct a detailed examination of the genital area with a magnifying glass. A blood and urine sample will be collected to test for infection. Each participant will use both the microbicidal gel and a placebo (contains no active ingredient) gel at different times during the study, and the results will be compared. Volunteers will participate up to 8 weeks.

DETAILED DESCRIPTION:
In Kenya, the HIV/AIDS epidemic has significantly increased adult and child mortality. Current prevention options, including the ABC model (Abstinence, Be faithful and correct and consistent Condom use) have not been sufficient to curb the generalized HIV epidemic. The development of topical microbicides provides a potential new prevention option against sexually transmitted infections (STIs), including HIV. Despite widespread use of topical microbicides among U.S. servicemen during World Wars I & II to prevent STI, the current HIV agenda has thus far focused almost exclusively on microbicide research for intravaginal use by females. Research on use of topical microbicides on the male genitalia has only examined potential adverse effects on the penis of microbicides intended for intravaginal or rectal use. Further research is necessary to determine what formulations, what doses, and what types of topical antimicrobials might prove acceptable, and tolerable for external genital use by male sub-populations, and effective for preventing HIV/STI in men. This Phase 1 safety trial is the culmination of a stepwise series of studies examining male genital hygiene and safety and acceptance of an alcohol-based topical microbicide among Kenyan men. The purpose of this randomized, double-blinded, placebo-controlled, crossover trial is to assess the safety and acceptability of 62% ethanol in emollient gel (intervention) and 15% ethanol in emollient gel (placebo), applied to the penis by men each morning and after every sexual exposure. The study population will include 30 healthy, uncircumcised Kenyan men working in the fishing industry. Participants will be randomly assigned to initial use of 1 of the 2 products for a 2-week interval. After a subsequent 2-week wash out period in which no topical gel will be used, the men will then cross over to use of the second product. The primary study objective is to assess the safety and toxicity of 62% and 15% ethanol in emollient gel on the penile epithelium and urethral mucosa. The secondary study objective is to assess the acceptability and compliance with the topical microbicide (62% ethanol) and placebo (15% ethanol) by men each morning and after each act of sexual intercourse. The primary study outcome measures include: self-reported urethral pain, urethral burning, penile itching, penile rash, penile blisters, penile ulceration or penile discharge at follow-up clinic visits on days 7, 14, 28, 35, 42 or 56; erythema (with or without induration), vesiculation, bullous reaction, and ulceration, of the penile shaft, foreskin, and glans, as observed by visual exam at follow-up clinic visits on days 7, 14, 28, 35, 42, or 56; erythema or ulceration of the urethral meatus, as observed by visual exam at follow-up clinic visits on days 7, 14, 28, 35, 42 or 56; and adverse events other than those listed as primary endpoints judged related to product use. The secondary study outcome measures are reported positive attributes (ease of use, increased pleasure during sex, positive feedback from primary sex partner) or negative attributes (difficulty of use, decreased pleasure during sex, negative feedback from primary sex partner) of the study products; reported willingness to use and recommend the products; and reported adherence with use of condoms and of the topical microbicide. Each participant will take part in the study for up to 8 weeks, including the screening period. The entire study should be completed within 5-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Working in the fishing industry for at least 3 months and living and working along the shores of Lake Victoria within a 70km radius of Kisumu, Kenya
* Uncircumcised
* Sexually active (have had sex in the last 2 weeks)
* Commercial or transactional sex during the past month
* Inconsistent condom use (less than 25% of all sex acts)
* Ability & willing to attend the clinic for a eight week period

Exclusion Criteria:

* STI diagnosis on clinical examination
* History of or evidence of dermatological inflammation (e.g. balanitis, phimosis, swelling of prepuce, warts on penis) upon clinical examination
* History of genital ulcer disease, penile trauma, dyspareunia (pain during sex), foreskin tears
* Congenital abnormalities: hypospadias, epispadias
* HIV, HSV-2 and syphilis-seropositive
* LE positive
* History of allergic reaction to alcohol products.
* Preference for oral sex
* Participating in HIV/HSV-2 or participated male circumcision studies based in Kisumu
* Investigator discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Self-reported urethral pain, urethral burning, penile itching, penile rash, penile blisters, penile ulceration or penile discharge. | At follow-up clinic visits on days 7, 14, 28, 35, 42 or 56.
Adverse events other than those listed as primary endpoints judged related to product use. | Varies

SECONDARY OUTCOMES:
Reported positive attributes or negative attributes of the study products, willingness to use and recommend the products, adherence with use of condoms and of the topical microbicide. | Varies

CONTACTS AND LOCATIONS:
Overall Officials: King K Holmes, MD, PhD, Principal Investigator — University of Washington; Elizabeth Bukusi, MBChB, MPH, PhD, Study Director — Kenya Medical Research Institute/University of Washington
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya